CLINICAL TRIAL: NCT06113562
Title: Patent Foramen Ovale Closure on Newly Diagnosed Patients With Obstructive Sleep Apnea and Refractory Hypoxia: A Pilot Study
Brief Title: Close Obstructive Sleep Apnea (OSA) Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn (Not able to enroll patients.)
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Eduardo De Marchena, Professor of Medicine and surgery, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20181090
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea; Patent Foramen Ovale
MeSH Terms: conditions — Sleep Apnea, Obstructive; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Persistent hypoxemia after Obstructive sleep apnea group (Experimental): Participants will receive Patent Foramen Ovale (PFO) closure and followed until repeat sleep apnea testing up to 6 months.
  Interventions: Procedure: PFO closure

INTERVENTIONS:
Procedure: PFO closure — The participants will receive a onetime closure of a small hole in heart. The procedure usually takes up to an hour. The procedure is done with local anesthesia and conscious sedation. A catheter is inserted into a vein in upper thigh and threaded to heart to deploy the closure device. Either Gore septal occluder or Amplatzer PFO occluder

SUMMARY:
The aim of this study is to evaluate the benefits of patent foramen ovale (PFO) closure on patients with obstructive sleep apnea (OSA) and persistent hypoxia despite optimal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with severe OSA, defined as an apnea-hypopnea index (AHI) greater than 30, associated with nocturnal saturation below 90%, as determined by a sleep medicine specialist using polysomnography.
2. Individuals need to have a patent foramen ovale documented by echocardiography.

Exclusion Criteria:

1. Individuals unable to take aspirin, clopidogrel, and/or ticagrelor.
2. Pregnant individuals or those who become pregnant during the course of the study will be automatically withdrawn.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
changes in the apnea hypoxia index | baseline and then up to 3 months after the study
  The Apnea hypopnea index that ranges from:
  0 to 5 is normal 5 to15 is mild 15 to 30 is moderate greater than 30 is severe.
change in mean nocturnal oxygen saturation | baseline and then up to 3 months after the study
  Oxygen saturation will be measured in percentage. Ranges from 0 to 100 percent. The higher the percent the higher the oxygen saturation.
change in duration of nocturnal oxygen desaturation duration. | baseline and then up to 3 months after the study
  Will be measured in seconds.

SECONDARY OUTCOMES:
change in quality of life as measured by the patient global impression of change scale. | baseline and then up to 3 months after the study
  Change Scale: Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
change in quality of sleep as measured by the Epworth Sleepiness Scale | baseline and then up to 3 months after the study
  Epworth Sleepiness Scale: The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing.
Change in physical activity as measured by Godin Leisure time physical activity questionnaire. | baseline and then up to 3 months after the study
  Self-reported leisure time physical activity as assessed by the Godin Leisure time physical activity questionnaire in all participants. Score range from 0 upwards, with higher scores indicating more leisure time physical activity.
change in fatigue as measured by the Fatigue Severity Scale. | baseline and then up to 3 months after the study
  Each item is scored between 1 and 7 (1 = strongly disagree, 7 = totally agree) in the scale consisting of 9 items that can be applied by individuals in a simple way. The total score range of the scale is 9-63. The total score is calculated by taking the average of 9 items. Accordingly, the lowest average score to be obtained is 1, and the highest average score is 7. The cut-off value was set at 4 and above to diagnose pathological fatigue. The lower the total score, the less fatigue.
changes in functional independence measure | baseline and then up to 3 months after the study
  The Functional independence measure (FIM) is an 18-item instrument comprising 13 motor items and 5 cognitive items, with each item graded on a 7-point ordinal scale (1 denotes complete dependence and 7 denotes complete independence), including the ability to perform activities of daily living (ADLs) across 6 areas (self-care, sphincter control, transfers, locomotion, communication, and social cognition). Total admission FIM (Ta-FIM) scores, total discharge FIM (Td-FIM) scores (18 - 126), motor FIM (m-FIM) sub-scores (13 - 91) and cognitive FIM (c-FIM) sub-scores (5 - 35), were tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo de Marchena, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No